CLINICAL TRIAL: NCT06459245
Title: Resistance Training to Prevent Lymphedema After Breast Cancer Surgery Randomized Controlled Study
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Yue WANG (Other)
Responsible Party: Sponsor-Investigator, Yue WANG, Yue WANG Deputy director, Peking University First Hospital
Organization: Peking University First Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023SF23
Record Dates: First submitted 2024-06-10; First posted 2024-06-14 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2024-06

CONDITIONS: Breast Cancer Female
Keywords: Breast cancer; resistance training; lymphedema; randomized control
MeSH Terms: conditions — Breast Neoplasms; Lymphedema | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine rehabilitation training (No Intervention): Starting from the first day after surgery, progressive progress was carried out according to the functional exercise table of the affected limb in the ward Functional exercise of affected limb; Pneumatic pressure pump physiotherapy during hospitalization: once a day, 30min each time;
- Resistance training (Experimental): Bend the dumbbell, hold a dumbbell in each hand, put it on the side of the body, bend the arm to lift the dumbbell, the front wall and the upper arm as close as possible; Hold the dumbbells flat on the side, with the back straight, stand with feet, arms perpendicular to the side of the body, hold the dumbbells with both hands, and lift the dumbbells to the side above shoulder level, elbows slightly bent; Stand with your feet straight, hold the dumbbells, and extend your arms back as far as possible. You can feel your upper arms and lower back being stretched. With your feet open, hold the dumbbells with both hands and extend your arms naturally in front of you. Lift them up until your elbows are above shoulder height and hold for 1-2 seconds.The training frequency is 2 to 3 times a week, 2 to 3 sets each time
  Interventions: Behavioral: Resistance training

INTERVENTIONS:
Behavioral: Resistance training — Bend the dumbbell, holding one dumbbell in each hand, on the side of the body, bend the arm to lift the dumbbell, front wall and upper arm as close as possible, pause for a moment, and then slowly lower the dumbbell until both arms are completely straight The second section of the dumbbell side flat, straight back, feet standing, arms perpendicular to the side of the body, hands grasp the dumbbell, to the side above the shoulder level, elbow slightly bent, and then put back in place The third section of the dumbbell rowing, feet stand straight, hold the dumbbell, the arm as far back as possible, can feel the upper arm and the waist back is stretched, and then straight back into the preparatory position Section 4: Lift the dumbbell flat in front of you, with your feet open, hold the dumbbell with both hands, extend your arms naturally in front of you, lift the dumbbell to the elbow above shoulder height, stay for 1-2 seconds.
  Arms: Resistance training

SUMMARY:
Breast cancer-related lymphedema is one of the most common chronic complications of breast cancer survivors. In existing studies, the reported incidence of lymphedema ranges from 2.5% to 42.9% . At present, there is no cure for lymphedema. Resistance training has been proved by many studies to alleviate the symptoms of lymphedema, improve the muscle strength of the upper limbs of patients, and improve the quality of life of patients, while not worsening lymphedema. Based on the best evidence, this study intends to construct resistance appropriate for this clinical scenario Training program: Conduct 3-month intervention for patients after breast cancer surgery to explore the effect of resistance training on the grip strength of the affected limb, the range of motion of the shoulder joint of the affected limb, the occurrence of lymphedema of the affected limb, quality of life, etc.

ELIGIBILITY:
Inclusion Criteria:

It was first diagnosed as grade I to III unilateral breast cancer by pathological examination； Breast cancer surgery was completed and axillary lymph node dissection was performed; To receive postoperative adjuvant treatment and follow-up in the outer fourth ward; Be able to communicate and exchange normally; Volunteer to participate in this research

Exclusion Criteria:

Extreme fatigue, severe anemia, ataxia, etc.; The presence of upper limb or shoulder problems from breast cancer treatment; Edema is in a non-stable stage (stable stage of edema means no treatment for edema in the past 3 months; No inflammation of the upper extremities requiring anti-infective treatment; No change in daily activities; Limb circumference change < 10%) ； Limited limb movement due to trauma, shoulder periarthritis, etc.; Limb braking is required for health reasons. Patients are lost to follow-up

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2025-06-24 (Estimated)

PRIMARY OUTCOMES:
Lymphedema occurrence | 3 months after intervention
  Tissue and local edema due to obstruction of lymphatic drainage

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No